CLINICAL TRIAL: NCT07138209
Title: A Phase 3 Randomized Study Comparing QLS32015 Monotherapy Versus Pomalidomide, Dexamethasone (Pd) or Selinexor, Dexamethasone (Sd) in Participants With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study Comparing QLS32015 Monotherapy Versus Pomalidomide, Dexamethasone (Pd) or Selinexor, Dexamethasone (Sd) in Participants With Relapsed or Refractory Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLS32015-301
Record Dates: First submitted 2025-08-13; First posted 2025-08-22 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — pomalidomide; selinexor; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLS32015 (Experimental): Participants will receive teclistamab monotherapy.
  Interventions: Drug: QLS32015
- Pomalidomide, Dexamethasone (Pd) or Selinexor and Dexamethasone (Sd) (Experimental): Participants will receive either Pd or Sd based on principal investigator's choice.
  Interventions: Drug: Pomalidomide; Drug: Selinexor; Drug: Dexamethasone

INTERVENTIONS:
Drug: QLS32015 — QLS32015 will be administered subcutaneously.
  Arms: QLS32015
Drug: Pomalidomide — Pomalidomide will be administered orally.
  Arms: Pomalidomide, Dexamethasone (Pd) or Selinexor and Dexamethasone (Sd)
Drug: Selinexor — Selinexor will be administered orally.
  Arms: Pomalidomide, Dexamethasone (Pd) or Selinexor and Dexamethasone (Sd)
Drug: Dexamethasone — Dexamethasone will be administered orally
  Arms: Pomalidomide, Dexamethasone (Pd) or Selinexor and Dexamethasone (Sd)

SUMMARY:
The purpose of this study is to compare the safety and efficacy of QLS32015 with Pd/Sd for the treatment of relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, regardless of gender.
* Subjects should be willing and able to comply with the study schedule and protocols.
* Documented initial diagnosis of multiple myeloma according to International Myeloma Working Group (IMWG) diagnostic criteria.Must have measurable disease as defined by the following: Serum M-protein greater than or equal to 1 g/dL; OR Urine M-protein greater than or equal to 200 mg/24 hours; OR Serum free light chain (FLC) assay; involved FLC level greater than or equal to 10 mg/dL provided the serum FLC ratio is abnormal.
* Received at least 3 prior lines of therapy, including a proteasome inhibitor (PI), an immunomodulatory drug, and an anti-CD38 monoclonal antibody (mAb).

Exclusion Criteria:

* Known hypersensitivity to any of the ingredients of this product.
* Diagnosis of active plasma cell leukemia or systemic light chain amyloidosis.
* Has any active severe mental illness, medical illness, or other symptoms/conditions that may affect treatment, compliance, or the ability to provide informed consent, as determined by the investigator.
* Disease is considered refractory to pomalidomide and selinexor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to 4 years
  PFS is defined as the time from the date of randomization to the date of first documented disease progression, as defined in the International myeloma working group (IMWG) 2016 response criteria, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Response (Partial Response [PR] or Better) | Up to 4 years
  Overall response (PR or better) is defined as participants who have a PR or better prior to subsequent antimyeloma therapy in accordance with the IMWG 2016 criteria.
Very Good Partial Response (VGPR) or Better Response | Up to 4 years
  VGPR or better (Stringent Complete Response [sCR]+Complete Response [CR]+VGPR) is defined as participants who achieve a VGPR or better response prior to subsequent antimyeloma therapy in accordance with the IMWG 2016 criteria.
Complete Response (CR) or Better Response | Up to 4 years
  CR or better response is defined as participants who achieve a CR or better response prior to subsequent antimyeloma therapy in accordance with the IMWG 2016 criteria
Duration of Response (DOR) | Up to 4 years
  DOR is defined as the time interval between the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease according to the IMWG 2016 response criteria or death due to any cause, whichever
Minimal Residual Disease (MRD) Negativity | Up to approximately 4 years
  MRD negativity is defined as participants who achieve MRD negativity at a threshold of 10^-5 at any timepoint after the date of randomization and before disease progression or start of subsequent antimyeloma therapy
Number of Participants with Adverse Events (AEs) by Severity | Up to 4 years
  Number of participants with AEs by Severity will be reported.
Change from Baseline in Symptoms, Functioning, and Overall Health-related Quality of Life (HRQoL) as Assessed by European Organization for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC-QLQ-C30) | Baseline up to 4 years
  Change from baseline scores